CLINICAL TRIAL: NCT03905174
Title: A Randomised, Single Blind Study Assessing Radiological Outcomes for Massive Segmental Femoral Replacements Using Either Porous Collar or Porous Collar With HA or Porous Collar With HA and Autologous Stem Cells
Brief Title: Massive Implants the Next Generation
Acronym: MING
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Iva Hauptmannova (Other)
Collaborators: Adler Ortho (Unknown)
Responsible Party: Sponsor-Investigator, Iva Hauptmannova, Head of Research & Innovation, Royal National Orthopaedic Hospital NHS Trust
Organization: Royal National Orthopaedic Hospital NHS Trust (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2017/MING
Record Dates: First submitted 2019-01-30; First posted 2019-04-05 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Bone Cancer; Bone Diseases
Keywords: revision surgery
MeSH Terms: conditions — Bone Neoplasms; Bone Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard treatment (Active Comparator): A porous collar for either distal or proximal femoral replacements
  Interventions: Device: custom made device
- standard treatment + HA (Active Comparator): A porous collar with hydroxyapatite (HA) for either distal or proximal femoral replacements
  Interventions: Device: custom made device
- standard treatment + HA + autogenic cells (Active Comparator): A porous collar with hydroxyapatite (HA) and stem cells for either distal or proximal femoral replacements
  Interventions: Device: custom made device

INTERVENTIONS:
Device: custom made device — surgical intervention to place custom made orthopaedic device
  Other Names: custom orthopaedic implantable device

SUMMARY:
The study will review the use of massive segmental replacements in the femur, which have a porous collar with and without HA, and autologous stem cell augment. This is a randomised controlled trial.

DETAILED DESCRIPTION:
The current surgical treatment of bone cancer patients and revision limb salvage requires usage of massive endoprosthetic bone implants. The incidence of aseptic loosening is a major cause of prosthesis failure in these patients, exploring ways to reduce such failures would allow extending longevity of massive implants in a relatively young population.

Current published literature stipulates that osteointegration could improve longevity of massive implants. Evidence suggests that usage of osteointegrated hydroxyapatite (HA) coated collar would reduce the incidence of aseptic loosening around the cemented intramedullary stem in distal femoral bone prosthesis

ELIGIBILITY:
Inclusion Criteria:

* Bone cancer patients requiring primary or revision femoral segmental replacements and non-cancer patients requiring revision femoral segment replacement for aseptic loosening
* Male or female, aged 18 years or above
* Able to provide consent

Exclusion Criteria:

* unable/unwilling to consent
* revisions surgery due to infection
* bone cancer patients excluded from stem cell arm
* bone cancer patients with pathological fractures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-09-20 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Radiological outcomes (X-ray, CT) | at 26 weeks (+/- 2 weeks)
  radiological outcomes to determine integration of implant into bone - bone growth
Radiological outcomes (X-ray, CT) | at 1 year (+/- 2 weeks)
  radiological outcomes to determine integration of implant into bone - bone growth
Radiological outcomes (X-ray, CT) | at 2 years (+/- 2 weeks)
  radiological outcomes to determine integration of implant into bone - bone growth

SECONDARY OUTCOMES:
Visual Analogue Score (VAS) pain score | up to 2 years (+/- 2 weeks)
  visual analogue pain score to determine improvement of pain over time, 0 to 10 scale will be used (0 = no pain, higher the number the worse the pain)

CONTACTS AND LOCATIONS:
Overall Officials: Panos Gikas, PhD FRCS, Principal Investigator — Royal National Orthopaedic Hospital NHS Trust
Locations (1):
- Royal National Orthopaedic Hospital NHS Trust, London, Middx, United Kingdom